CLINICAL TRIAL: NCT03550742
Title: Real-World Perception of Tolerability and Bowel Function Effects of Fuco-N-Tetraose in IBS Patients
Brief Title: Effect of HMOs as Nutritional Support for Normal Bowel Movements in IBS Patients
Acronym: GRIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycom, Inc. (Industry)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor
Organization: Glycom A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GRIPS; CT-2017-01 (Other: IntegReview IRB)
Record Dates: First submitted 2018-05-09; First posted 2018-06-08 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Human Milk Oligosaccharides; IBS-C; IBS-D; IBS-M
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Daily administration of 5g of Fuco-N-Tetraose as a bolus for a period of 12 weeks.
  Interventions: Other: Fuco-N-Tetraose

INTERVENTIONS:
Other: Fuco-N-Tetraose — Daily bolus of Fuco-N-Tetraose

SUMMARY:
This is an open labeled, one-armed real-world study in IBS-patients. All participants will receive active treatment for 12 weeks.

The primary objective of the study is to assess the effect of Human Milk Oligosaccharides (HMOs) on bowel function in adults with IBS. Secondary objectives are to evaluate HMOs' tolerability, effect on participant reported satisfaction with bowel habits, interference with life in general, quality of life, somatic symptoms, and anxiety and depression in all patients and subgroups of patients.

DETAILED DESCRIPTION:
In this trial, a total of 300 adults (at least 18 years of age) diagnosed with irritable bowel syndrome (IBS) in accordance with the Rome IV criteria will be included. Patients will be recruited from gastroenterologists and primary care clinics across the USA. The study product, Fuco-N-Tetraose, will be taken daily throughout the course of the trial. All data will be collected through 4 web based surveys, and the participants will complete those at baseline before the intervention starts, and after 4, 8 and 12 weeks of intake of the study product.

The primary outcome of the study will be assessed by the Patients' Global Impression of Change (PGIC) scale. Other questionnaires used in the study includes the IBS specific Gastrointestinal Symptom Rating Scale (GSRS-IBS), the IBS Quality of Life Scale (IBS-QoL), the Participant Health Questionnaire-4 (PHQ-4), the Participant Health Questionnaire-12 (PHQ-12), and the Bristol Stool Form Scale (BSFS). All outcomes will be evaluated in all patients and in sub-groups of patients. i.e. subtypes by predominant bowel habit (diarrhea-predominant, constipation-predominant, or altered/mixed pattern), and lactose intolerant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give oral and written informed consent
2. Age minimum 18 years at enrolment
3. Current clinical diagnosis of IBS from a healthcare provider, and meeting Rome IV IBS diagnostic criteria
4. Ability and willingness to understand and comply with the study procedures
5. Ability to read, speak and understand English
6. Free access to the internet via computer, tablet or smartphone to complete study surveys and also to allow for study team follow-up as needed.

Exclusion Criteria:

1. Participation in a clinical intervention study one month prior to screening visit and throughout the study.
2. Medically diagnosed with celiac disease, Crohn's disease, ulcerative colitis, diverticulitis, inflammatory bowel disease, or clostridium difficile infection by a doctor
3. Pregnant or lactating or wish to become pregnant during the period of the study.
4. Lack of suitability for participation in the study for any reason as judged by the site investigator or Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in bowel function | Baseline and after 4, 8 and 12 weeks of intake
  Change from baseline in bowel function assessed as the proportion of bowel movements with abnormal fecal consistency measured with the Bristol Stool Form Scale

SECONDARY OUTCOMES:
Change in patients' perception of body function | Baseline and after 4, 8 and 12 weeks of intake
  Change from baseline in patients' perception of body function measured by the Patients' Global Impression of Change (PGIC) scale.
Evaluate tolerability of fuco-N-tetraose | Baseline and after 4, 8 and 12 weeks of intake
  Evaluate tolerability of fuco-N-tetraose using GSRS-IBS
Evaluate tolerability of fuco-N-tetraose | Baseline and after 4, 8 and 12 weeks of intake
  Evaluate tolerability of fuco-N-tetraose using IBS-SSS
Change in satisfaction with bowel habits | Baseline and after 4, 8 and 12 weeks of intake
  Change from baseline in satisfaction with bowel habits measured with IBS-SSS
Change in IBS' interference in life in general | Baseline and after 4, 8 and 12 weeks of intake
  Change from baseline in IBS' interference in life in general measured with IBS-SSS
Change in quality of life | Baseline and after 4, 8 and 12 weeks of intake
  Change from baseline in quality of life measured with the IBS Quality of Life Scale (IBS-QoL)
Change on somatic symptoms | Baseline and after 4, 8 and 12 weeks of intake
  Change from baseline on somatic symptoms measured with the Participant Health Questionnaire-12 (PHQ-12)
Change in anxiety and depression | Baseline and after 4, 8 and 12 weeks of intake
  Change from baseline in anxiety and depression measured with the Participant Health Questionnaire-4 (PHQ-4)

CONTACTS AND LOCATIONS:
Overall Officials: Olafur Palsson, PsyD, Prof, Principal Investigator — UNC-Chapel Hill School of Medicine
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palsson OS, Peery A, Seitzberg D, Amundsen ID, McConnell B, Simren M. Human Milk Oligosaccharides Support Normal Bowel Function and Improve Symptoms of Irritable Bowel Syndrome: A Multicenter, Open-Label Trial. Clin Transl Gastroenterol. 2020 Dec;11(12):e00276. doi: 10.14309/ctg.0000000000000276. PMID 33512807